CLINICAL TRIAL: NCT03047863
Title: The Therapeutic Effect of Topical EGF Cream for Dermatologic Adverse Events Related to EGFR Inhibitors
Brief Title: Therapeutic Effect of EGF Cream for Cutaneous Adverse Event of EGFR Inhibitors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VC16EISI0179
Record Dates: First submitted 2016-12-02; First posted 2017-02-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Epidermal Growth Factor
Keywords: Epidermal Growth Factor
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repair Control EGF® (Experimental): EGF cream was applied. Half of face was treated with emollient containing EGF.
  Interventions: Drug: Repair Control EGF®
- Cream without rhEGF (Placebo Comparator): Placebo cream without EGF was applied. The other half of face was treated with only emollient which was not containing EGF.
  Interventions: Drug: Cream without rhEGF

INTERVENTIONS:
Drug: Repair Control EGF® — A Split face study was done. Patients applied 1 finger tip unit of EGF cream on one side of face, twice a day for 4 weeks.
  EGF cream(Repair Control EGF®) containing 10 ppm of rhEGF was prepared at D.N. Co., Ltd. (Seoul, South Korea)
  Other Names: EGF cream containing 10 ppm of rhEGF
  Arms: Repair Control EGF®
Drug: Cream without rhEGF — A Split face study was done. Patients applied 1 finger tip unit of cream on the other side of face, twice a day for 4 weeks.
  Placebo cream was prepared at at D.N. Co., Ltd. (Seoul, South Korea), consisted of same ingredient with EGF cream except rhEGF
  Arms: Cream without rhEGF

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of topical EGF cream for dermatologic adverse events related to EGFR inhibitors.

DETAILED DESCRIPTION:
Epidermal growth factor receptor(EGFR) is involved in cell proliferation and is overexpressed or abnormally activated in malignant tumors originating from the colon, breast, ovary, pancreas, and lung. EGFR tyrosine kinase inhibitor(TKI), gefitinib, erlotinib, and afatinib have been for the treatment of cancer associated with EGFR gene mutation. In addition, monoclonal antibodies to EGFR, such as cetuximab and panitumumab, have been used as a chemotherapy for rectal cancer without ras gene mutation and advanced head and neck cancer.

The incidence of cutaneous toxicity of EGFR inhibitors is reported to be 75-80%. Clinical features include acneform folliculitis, xerosis, paronychia, and itching. Of these, about 10% of patients with Grade 3 or greater have a detrimental effect on quality of life and adherence to treatment, resulting in impaired therapeutic results.

There have been many attempts to prevent or treat such skin toxicity. However, there has been no scientifically proven treatment until now.

There is a growing interest in the role of EGF emulsifiers in the treatment of skin adverse effects of EGFR inhibitors, as a result of studies that improve acne significantly compared to placebo.

The purpose of this study is to evaluate the therapeutic efficacy of EGF cream in the treatment of skin adverse effects in patients with malignant tumors treated with EGFR inhibitor (TKI or monoclonal antibody).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received EGFR inhibitors (gefitinib, erlotinib, afatinib, cetuximab, etc.) for malignant tumors
* Patients with EGFR inhibitor-associated skin reactions: National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE V4.03) Grade 2, 3 Patients
* Patients who can understand and follow the protocol
* Patients who spontaneously agreed to the study

Exclusion Criteria:

* NCI-CTCAE grade 4 patients requiring systemic drug therapy
* Those with a history of antibiotic treatment, local and systemic steroid therapy within 4 weeks for reasons other than EGFR inhibitors
* Patients with existing acne history
* Patients who have already received anti-EGFR therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of severity of acneform eruption induced by EGFR inhibitors | Baseline, 1 week, 2 weeks, 4 weeks
  To evaluate the severity of acneiform eruption, the investigators take a photograph of full face. The number of inflammatory and noninflammatory lesions will be counted and accessed the severity based on the Korean Acne Grading System(KAGS).

SECONDARY OUTCOMES:
change of skin hydration | Baseline, 1 week, 2 weeks, 4 weeks
  Skin hydration is measured with Corneometer® (CM820/825; C-K Electronics, Cologne, Germany).
  It shows the skin moisturizing condition in arbitrary units(AU) and the unit is from 0 to 220.
change of sebum production | Baseline, 1 week, 2 weeks, 4 weeks
  Sebum production is measured with Sebumeter® (SM815; C-K Electronics, Cologne, Germany).
  It measured at forehead, cheek and chin, presented as ㎍/㎠.
Investigator's global assessment score | Baseline, 1 week, 2 weeks, 4 weeks
  Investigator's global assessment (IGA) Score : It will be assessed as a 5-point scale (-1 = worsen, to 3 = marked improvement).
Patient's global assessment score | Baseline, 1 week, 2 weeks, 4 weeks
  Patient's global assessment (PGA) score will be assessed as a 5-point scale (-1 = worsen, to 3 =marked improvement).
The side effects of product | Baseline, 1 week, 2 weeks, 4 weeks
  It will be assessed by patient-report.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Bae, MD, PhD, Study Chair — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided